CLINICAL TRIAL: NCT01336543
Title: A Pilot Study: Phase II Study of Histology-based Consolidation Chemotherapy Following Concurrent Chemo-radiotherapy for Inoperable Stage III Non-small Cell Lung Cancer
Brief Title: Consolidation Chemotherapy/Concurrent Chemo-radiotherapy for Inoperable Stage III Non-small Cell Lung Cancer (NSCLC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual, small patient population at center.
Sponsor: Syed Jafri (Other)
Responsible Party: Sponsor-Investigator, Syed Jafri, Assistant Professor, Louisiana State University Health Sciences Center Shreveport
Organization: Louisiana State University Health Sciences Center Shreveport (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H11-071
Record Dates: First submitted 2011-04-12; First posted 2011-04-18 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Stage III Non-small Cell Lung Cancer
Keywords: Non small cell lung cancer; Inoperable Stage III; Inoperable; Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Gemcitabine; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active Treatment (Experimental): ACTIVE TREATMENT intervention below:
  1. NSCLC (Non-Small Cell Lung Cancer)
  2. PE (Cisplatin 50mg/m2 on days 1,8,29,36 Etoposide 60 mg/m2 days 1-3 and 29-31)
  3. Radiation 59.4 Gy with 2 cycles of PE
  4. (Non-squamous histology) Pemetrexed consolidation 500mg/m2 every 21 days for 4 cycles
  5. (Squamous histology) Gemcitabine consolidation 1000mg/m2 days 1,8, every 21 days for 4 cycles
  Interventions: Drug: Chemotherapy following concurrent Chemoradiotherapy

INTERVENTIONS:
Drug: Chemotherapy following concurrent Chemoradiotherapy — 1. NSCLC (Non-Small Cell Lung Cancer)
  2. PE (Cisplatin 50mg/m2 on days 1,8,29,36 Etoposide 80mg/m2 days 1-3 and 29-31)
  3. Radiation 59.4 Gy with 2 cycles of PE
  4. (Non-squamous histology) Pemetrexed consolidation 500mg/m2 every 21 days for 4 cycles
  5. (Squamous histology) Gemcitabine consolidation 1000mg/m2 days 1,8, every 21 days for 4 cycles
  Other Names: Pemetrexed; Gemcitabine; Cisplatin; Etoposide

SUMMARY:
This is a pilot phase II study of histology based consolidation chemotherapy in patients with inoperable stage III Non-Small Cell Lung Cancer (NSCLC) following concurrent chemo-radiotherapy. Patients with inoperable stage III NSCLC would be treated with standard concurrent chemo-radiotherapy and subsequently those with non-squamous histology would be offered 4 cycles of consolidation pemetrexed and those with squamous histology 4 cycles of consolidation with gemcitabine.

DETAILED DESCRIPTION:
Non-Small Cell Lung Cancer (NSCLC) is the leading cause of cancer related mortality in US (1). About 22% of patients diagnosed with NSCLC have locally advanced or stage III disease at the time of diagnosis (2). 5 years survival for stage III lung cancer is 23% which is much less than survival in similar stage breast and Colon Cancers (2). Current standard of care for inoperable stage III NSCLC is concurrent chemo-radiotherapy as established by a study (Southwestern Oncology Group) SWOG 9019 (3). Surgery following concurrent chemo-radiotherapy has been evaluated in a large Phase III clinical trial in patients with Stage III (N2) disease which did not show any improvement in overall survival from surgery as compared to concurrent chemo-radiotherapy alone.(4). These two studies demonstrated that the most common site of cancer relapse in patients with stage III disease was distant metastasis, 65% (3) and 57% (4) respectively.

These observations have led to the idea that perhaps giving additional chemotherapy following definitive concurrent chemo-radiotherapy may prevent distant relapse in stage III NSCLC.

This idea was evaluated in a Phase II study SWOG S9504 in which patients with stage III NSCLC were treated with concurrent chemo-radiotherapy followed by 4 cycles of docetaxel consolidation (5). Four cycles of docetaxel consolidation showed an impressive improvement in median Overall Survival (OS) to 26 months.

This idea of docetaxel consolidation was subsequently evaluated in a large phase III trial in which patients inoperable stage III NSCLC after receiving concurrent chemo-radiotherapy were randomized to docetaxel consolidation versus observation (6). However, this study showed no improvement in OS between the docetaxel arm and the observation arm. Many patients in docetaxel arm developed pneumonitis and febrile neutropenia.

Histology based selection of chemotherapy is now standard of for stage IV metastatic NSCLC. A large randomized Phase III trial from Europe showed that a combination of Cisplatin and Pemetrexed is more effective in patients with non-squamous histology and a combination of Cisplatin and Gemcitabine showed efficacy in patients with squamous cell histology (7). Recently maintenance Pemetrexed was evaluated in advanced NSCLC and showed improvement in PFS and OS in patients with non-squamous histology (8). Similarly maintenance gemcitabine has also been evaluated in large Phase III clinical trial after initial chemotherapy with Cisplatin and Gemcitabine (9).

Since most patients with inoperable stage III NSCLC develop distant metastasis following definitive concurrent chemo-radiotherapy there clearly is a need to give addition treatment for these patients. Docetaxel consolidation has not been shown to be successful as noted above. Perhaps tailoring chemotherapy according to histology may result in improvement in PFS and OS in these patients.

Based on this hypothesis the investigators intend to do a pilot phase II study of histology based consolidation chemotherapy in patients with inoperable stage III NSCLC following concurrent chemo-radiotherapy. Patients with inoperable stage III NSCLC would be treated with standard concurrent chemo-radiotherapy and subsequently those with non-squamous histology would be offered 4 cycles of consolidation pemetrexed and those with squamous histology 4 cycles of consolidation with gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 18 years and older with histology proven NSCLC with inoperable stage III A or IIIB disease.
2. Inoperable stage III A defined by multiple and or/bulky N2 mediastinal lymph nodes on computed tomography (CT) scan such that in opinion of treating investigator, the patient was not a candidate for surgical resection.
3. N2 disease must be documented by either biopsy, fluorodeoxyglucose positron emission tomography (PET), and or CT scan if nodes are more than 2 cm.
4. Stage IIIB patients must have N3 or T4 status. N3 status must be documented by presence of contralateral (to the primary tumor) mediastinal lymph node or supraclavicular or scalene lymph node proven by either biopsy, fluorodeoxyglucose PET, or more than 2 cm on CT scan.
5. No prior treatment for lung cancer
6. ECOG Performance status of 0-1.
7. Initiation of consolidation chemotherapy within 4-8 weeks of concurrent chemo-radiotherapy without progression.
8. Adequate organ function

   * leukocytes >3,000/mcL
   * absolute neutrophil count >1,500/mcL
   * platelets >100,000/mcL
   * total bilirubin within normal institutional limits
   * AST (SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
   * creatinine within normal institutional limits OR
   * creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal

   All labs should be obtained within 14 days prior to start of study drug treatment.
9. Ability to give informed consent and willingness to adhere to study protocol.

Exclusion Criteria:

1. Patient who have had prior treatment for lung cancer.
2. Prior history of radiation to chest.
3. Known malignancy other than the current cancer.
4. Uncontrolled intercurrent illness including but not limited to ongoing active infection, history of cardiac disease, e.g. uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within last six months or ventricular arrhythmias requiring medication, psychiatric illness that would impair patients ability to comply with study requirements.
5. Pregnant or lactating women (any women becoming pregnant during the study will be withdrawn from the study)
6. Patient with documented or symptoms of peripheral neuropathy.
7. History of allergic reaction to compounds similar to the ones used in this study.
8. Malignant effusions (pleural or pericardial)
9. Superior sulcus (Pancoast) tumors.
10. Any condition that would hamper ability to give informed consent or ability to comply with study protocol.
11. HIV patients on anti-retroviral therapy are in-eligible to participate in this study because of potential interaction with the study drugs and increase susceptibility for infections during course of marrow suppressive chemotherapy and radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 3 years
  From date of registration to date of first observation of progressive disease, death due to any cause or symptomatic deterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Syed H. Jafri, MD, Principal Investigator — LSU Health Shreveport, Feist-Weiller Cancer Center
Locations (1):
- LSU Health Sciences Center, 1501 Kings Highway, Shreveport, Louisiana, United States